CLINICAL TRIAL: NCT07338448
Title: The Effect of Electrical Acupoint Stimulation on Gastric Reflux During Anesthesia With I-gel Ventilation
Brief Title: Electrical Acupoint Stimulation on Gastric Reflux During I-gel Ventilation
Acronym: ASGARD-igel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJH-A-20251021
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia
Keywords: acupoint stimulation; general anesthesia; gastric reflux; igel
MeSH Terms: conditions — Gastroesophageal Reflux; Ige Responsiveness, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical stimulation (Experimental): Electrodes are pasted at the Neiguan, Zusanli, Gongsun, Taichong acupoints and electrical stimulation is given from anesthesia induction to end of surgery
  Interventions: Other: transcutaneous electrical acupoint stimulation; Other: electrodes attachment
- Control (Placebo Comparator): Electrodes are pasted at the Neiguan, Zusanli, Gongsun, Taichong acupoints but no electrical stimulation is given
  Interventions: Other: electrodes attachment

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation — electrical stimulation at 2Hz/10Hz is given from induction to end of surgery
  Arms: Electrical stimulation
Other: electrodes attachment — Electrodes are pasted to the skin of Neiguan, Zusanli, Gongsun, Taichong acupoints

SUMMARY:
This study will compare the effects of transcutaneous acupoint electrical stimulation versus no stimulation on intraoperative gastric reflux in patients undergoing general anesthesia with i-gel airway device ventilation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* scheduled for surgery under general anesthesia with igel ventilation

Exclusion Criteria:

* American society of anesthesiologists status higher than grade 3
* history of gastrointestinal surgery
* Currently taking acidic medications, or medications that affect gastric acid secretion or gastrointestinal motility
* High risk of reflux or aspiration (e.g., symptomatic gastroesophageal reflux disease or hiatal hernia)
* History of postoperative nausea and vomiting (PONV)
* Intraoperative requirement of Trendelenburg position
* Expected surgery duration exceeding 4 hours
* Contraindications for acupoint electrical stimulation, such as patients with implanted electrophysiological devices, or skin infection/lesions at acupoint sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
pH value at middle-esophageal part at end of surgery | at end of surgery

SECONDARY OUTCOMES:
number of gastric reflux episodes | from intubation of igel to end of surgery, at an average of 2 hours
total duration of gastric reflux episodes | from intubation of igel to end of surgery, at an average of 2 hours
longest duration of gastric reflux episodes | from intubation of igel to end of surgery, at an average of 2 hours
pH value at glottis at the end of surgery | at end of surgery
percentage of patients suffering postoperative nausea and vomiting by 24 hours after surgery | from end of surgery to 24 hours after surgery

IPD SHARING:
Plan to Share IPD: Undecided